CLINICAL TRIAL: NCT01641289
Title: Paracetamol Effect on Oxidative Stress and Renal Function in Severe Falciparum Malaria With Intravascular Haemolysis: A Randomised Controlled Clinical Trial
Brief Title: Paracetamol Effect on Oxidative Stress and Renal Function in Severe Malaria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAKMAL1201
Record Dates: First submitted 2012-05-23; First posted 2012-07-16 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Malaria
Keywords: Falciparum malaria; Paracetamol; Renal function; Oxidative stress
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paracetamol (Experimental): >50kg: Paracetamol 1gm PO/NG q6hourly for 72 hours and febrile for 24 hours (maximum total dose 4g/24 hours) plus intravenous Artesunate
  <50kg: Paracetamol 12.5-15mg/kg/dose q6hourly for 72 hours and febrile for 24 hours (maximum total dose 5 doses/24hours;75mg/kg) plus intravenous Artesunate
  Interventions: Drug: Paracetamol
- No Paracetamol (Active Comparator): No paracetamol + Intravenous Artesunate
  * If temperature > 40°C, ibuprofen PO/PR will be administered in the absence of renal impairment and dehydration; 500mg paracetamol PO/PR will be administered in the presence of renal impairment or dehydration. Dengue testing will be done prior to the administration of ibuprofen.
  Interventions: Drug: No Paracetamol

INTERVENTIONS:
Drug: Paracetamol — >50kg: Paracetamol 1gm PO/NG q6hourly for 72hours and afebrile for 24h (maximum total dose 4g/24 hours) plus intravenous Artesunate <50kg: Paracetamol 12.5-15mg/kg/dose q6hourly for 72hours and afebrile for 24h (maximum total dose 5 doses/24hours;75mg/kg) plus intravenous Artesunate
  Arms: Paracetamol
Drug: No Paracetamol — No paracetamol + Intravenous Artesunate
  * If temperature > 40°C, ibuprofen PO/PR will be administered in the absence of renal impairment and dehydration; 500mg paracetamol PO/PR will be administered in the presence of renal impairment or dehydration. Dengue testing will be done prior to the administration of ibuprofen.
  Arms: No Paracetamol

SUMMARY:
Blackwater fever, characterized by intravascular haemolysis and hemoglobinuria, is an important cause of renal impairment and mortality in severe malaria caused by Plasmodium falciparum. The largest malaria clinical trials report blackwater incidences of 5-7% in Asian adults and 4% in African children with severe malaria treated with artesunate or quinine. The prevalence of blackwater fever in Chittagong, Bangladesh is 15% with associated rates of renal failure and mortality of 42.9% and 14.2% respectively.

The fundamental characteristic of blackwater fever is the presence of intravascular hemolysis of both infected and uninfected erythrocytes and release of free haemoglobin. The cytotoxic free haemoglobin present can cause severe oxidative damage as a result of haem redox cycling yielding ferric and ferryl heme, which generate radical species that induce lipid peroxidation and subsequent production of F2-isoprostanes (F2-IsoPs). Evidence suggests that F2-IsoPs generated by the hemoprotein-catalyzed oxidation of lipids are responsible for the oxidative damage and vasoconstriction associated with renal injury in haemolytic disorders and rhabdomyolysis.

A novel mechanism of paracetamol was recently demonstrated, showing that paracetamol is a potent inhibitor of hemoprotein-catalyzed lipid peroxidation by reducing ferryl heme to its less toxic ferric state and quenching globin radicals. In a recent proof of concept trial, paracetamol at therapeutic levels was shown to significantly decrease oxidant kidney injury, improve renal function and reduce renal damage by inhibiting the hemoprotein-catalyzed lipid peroxidation in a rat model of rhabdomyolysis-induced renal injury. Since adults with severe malaria demonstrate increased concentrations of cell-free haemoglobin, and urinary F2-IsoPs, the investigators hypothesize that this novel inhibitory mechanism of paracetamol may provide renal protection in this population by reducing the hemoprotein-induced lipid peroxidation. As there is currently no consensus that exists concerning adequate medical treatment for blackwater fever, the potential application of this safe and extensively used drug would be of great benefit.

DETAILED DESCRIPTION:
Mortality in severe malaria remains ~15% despite the best available parasiticidal antimalarial therapy, intravenous artesunate. Adjunctive therapies in combination with anti-parasitic drugs have the potential to improve outcomes. However, currently there are no proven adjunctive therapies for the treatment of severe malaria, which can improve case-fatality when used in combination with anti-parasitic drugs. This research proposal focuses on exploring if paracetamol prevents renal dysfunction caused by free haemoglobin induced oxidative damage in severe malaria.

Blackwater fever epidemiology As early as the 1800s, blackwater fever complicating severe malaria caused by Plasmodium falciparum was recognized as an important cause of morbidity and mortality, with a 25-30% mean mortality rate. The etiology and pathogenesis is poorly understood but it is characterized by massive intravascular haemolysis and passage of black or red urine, which can lead to renal impairment and death. This manifestation was linked to quinine therapy as its occurrence nearly disappeared during the chloroquine era from 1950 to 1980. Since 1990, the resurgence in the number of cases noted in both malaria-free and malarious areas in non-immune and immune individuals has generated renewed interest into this manifestation of severe malaria. The largest malaria clinical trials report blackwater fever incidences of 7% and 4% in Asian adult patients with severe malaria treated with artesunate and quinine, respectively and 4% in African children treated with either drug. The prevalence of blackwater fever in Chittagong, Bangladesh was recently determined in a pilot study to be 15% with associated renal failure and mortality rates of 42.9% and 14.2% respectively.

Blackwater fever pathogenesis Although the exact mechanism linking falciparum malaria and blackwater fever is uncertain, numerous explanations have been suggested. It has been proposed to occur in 4 specific circumstances: (1) in case patients with G6PD deficiency with or without malaria who take oxidant drugs (primaquine) (2) in case patients with G6PD deficiency and malaria untreated and treated with quinine (3) when patients (normal G6PD) with severe malaria are treated with quinine (4) when people exposed to malaria self-medicate with quinine or related amino-alcohol drugs. However, new circumstances of blackwater fever have emerged, occurring in patients with normal G6PD levels with severe malaria who have received artesunate rather than quinine.

Role of oxidative stress and free haem The fundamental characteristic of blackwater fever is the presence of massive haemolysis of both infected and uninfected erythrocytes and release of free haemoglobin. The free haem is highly cytotoxic, and an important scavenger of nitric oxide, promoting endothelial damage and is proposed to be involved in the pathogenesis of renal injury and cerebral malaria. When the degree of intravascular haemolysis exceeds the capacity of plasma haptoglobin to bind the haemoglobin released from red blood cells, free haemoglobin is then filtered by the glomeruli and enters the renal tubules. In a series of renal biopsies, fine and coarse haemoglobin granules are present in the proximal tubules, while haemoglobin casts and granular casts predominate in the distal and collecting tubules in patients with blackwater fever and intravascular haemolysis. This classic theory of renal damage by tubular precipitation is challenged by recent findings of reversing oxidative properties of free haem can prevent renal damage. The free haemoglobin present is pathogenic as the ferrous haem can be oxidized to the ferric state (FeIII) subsequently conferring peroxidase activity to the haemoglobin. Consequently, the haemoglobin can reduce hydroperoxides, such as hydrogen peroxide (H2O2) and lipid hydroperoxides, which generate the ferryl state (FeIV=O) of haemoglobin and a globin protein radical.

Haem Fe(III) protein + H2O2 --> haem [Fe(IV)=O] protein• + H+ + H2O The ferryl haem and protein radical can then generate lipid radicals by oxidation of free and phospholipid-esterified unsaturated fatty acids. The arachidonic side chains of membrane phospholipids are particularly vulnerable to this free radical-mediated damage in the complex cascade of lipid oxidation leading to the generation of F2-isoprostanes (F2-IsoPs) and isofurans (IsoFs). Evidence suggests that F2-isoPs generated by the haemoprotein-catalyzed oxidation of lipids are responsible for the oxidative damage and vasoconstriction associated with renal injury in the setting of hemolytic disorders and rhabdomyolysis.

Paracetamol and oxidative stress A novel mechanism of paracetamol was recently demonstrated, showing that paracetamol acts as a potent inhibitor of haemoprotein-catalyzed lipid peroxidation by reducing ferryl haem to its less toxic ferric state and quenching globin radicals. This effect is enhanced 14-fold in an acidic milieu. In a recent proof of concept trial, paracetamol at therapeutic levels was shown to significantly decrease oxidant injury in the kidney, improve renal function and reduce renal damage by inhibiting the haemoprotein-catalyzed lipid peroxidation, mediated by redox cycling of the haem moiety of myoglobin, in a rat model of rhabdomyolysis-induced renal injury.

Rationale Since adults with severe malaria and blackwater fever associated with haemolysis demonstrate increased concentrations of cell-free haemoglobin, severe acidosis and urinary F2-IsoPs, the investigators hypothesize that this novel inhibitory mechanism of paracetamol may provide renal protection in this population by reducing the haemoprotein-induced lipid peroxidation. As there is currently no consensus that exists concerning adequate medical treatment for blackwater fever, the potential application of this safe and extensively used drug would be of great benefit.

Proposed activities The main activity proposed is a randomised open label controlled study of paracetamol in patients with severe falciparum malaria to assess its modulating effect on renal function and oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age >12 years
2. Presence of severe or moderately severe P. falciparum malaria, with and without blackwater fever, confirmed by positive blood smear with asexual forms of P. falciparum
3. Temperature >38 degrees Celsius on admission or fever during the preceding 24hours
4. Written informed consent from patient or attending relative able to and willing to give informed consent. Consent form and information sheets will be translated into Bangla and copies provided to the patient.

Exclusion Criteria:

1. Patient or relatives unable or unwilling to give informed consent
2. History of chronic liver disease
3. History of alcohol use (>3drinks per day)
4. Contraindication or allergy to paracetamol or artesunate therapy
5. Contraindication to nasogastric tube insertion i.e. facial fracture, bleeding diathesis
6. Pregnancy

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-07-10 (Actual); Primary Completion 2014-09-13 (Actual); Study Completion 2014-09-21 (Actual)

PRIMARY OUTCOMES:
Effect of paracetamol concentrations | 72 hours
  Compare the effect of therapeutic paracetamol concentrations compared with absent or low paracetamol concentration on renal function, peak creatinine levels or trough creatinine clearance, defined as the change at 72 hours compared to baseline, in patients with severe and moderately severe falciparum malaria stratified by the level of intravascular haemolysis (cell-free haemoglobin).

SECONDARY OUTCOMES:
Compare treatment arm with control arm with respect to duration of Acute Kidney Injury (AKI) and development of AKI. | 14 days
  Duration of AKI will be defined as the length of time elapsed until serum creatinine returns to normal (<1mg/dL) in the absence of renal replacement therapy. Development of AKI will be assessed using the Acute Kidney Injury Network (AKIN) criteria, and by a creatinine increase of >= 0.5mg/dl or 25%. Plasma paracetamol concentration will be measured daily by liquid chromatography-mass spectrometer (LC-MS/MS).
Compare between groups correlations between oxidative stress, cell-free hemoglobin and renal function | 3 days
  Urine and plasma F2-isoprostanes and isofurans will be measured by gas chromatography-mass spectrometry. Cell-free haemoglobin measured as plasma concentration by enzyme linked immunosorbent assay (ELISA) on admission then daily for 72hours. Cell free haem measured in plasma using a chromogenic assay on admission then daily for 72hours. Haem-to-protein cross-links measured by high performance liquid chromatography (HPLC) on admission and daily for 72hours.
Assessment of Blackwater fever and association with renal function | 7 days
  Blackwater fever assessed using a standardized urine colour chart and urine haemoglobin every 6 hours until clinical recovery between groups.
Mortality and hemodialysis trends | 4 weeks
  To compare mortality and hemodialysis trends between groups and evaluate if they correlate with level of oxidative stress, cell free haemoglobin and renal function.
Host factors of Intravascular Haemolysis | 4 weeks
  Intravascular haemolysis according to G6PD status.
Fever clearance time | 7 days
  Compared fever clearance time defined as the time taken for the tympanic temperature to fall below 37.5°C and remain there for at least 24hours); Fever time defined as the duration in hours of an individuals temperature above 37.5°C; Area above the 37.5°C temperature versus time curve (AUC-T°) within first 24hours of treatment. Aural temperature will be measured every 6 hours until fever clearance.
Parasite clearance time | 7 days
  Parasite clearance time assessed by microscopy of peripheral blood films will be assessed every 6hours for the presence of asexual parasitaemia until negative on 2 consecutive blood films. Parasite half lives and clearance time will be compared between groups. Parasites will also be staged to assess if sequestration is inhibited due to temperature reduction.
Parasite sequestration | 7 days
  Parasite sequestration assessed by capillary flow in the rectal microcirculation using Orthogonal Polarization Spectral (OPS) imaging will be compared between groups.
Assessment of Acute Kidney Injury | 7 days
  Evaluation of pre-renal and acute tubular necrosis assessed by blood and urine biomarkers of pre-renal and renal injury including neutrophil gelatinase-associated lipocalcin (NGAL) and kidney injury molecule (KIM).
Urine scoring of dehydration and haemolysis | 72 hours
  Urine colour will be assessed by standardized urine colour charts. Urine colour will be correlated with urine specific gravity, urine osmolality, urine haemoglobin and creatinine clearance.
Safety assessment | 6 weeks
  Safety assessed by the number of patients with serious adverse events (SAEs) and by changes from baseline in vital signs and laboratory measurements.
Assess the antimalarial drug sensitivity of patients treated with paracetamol | 72 hours
  Preliminary in vitro studies suggest that paracetamol potentiates the anti-parasitic effect of artesunate as lower 50% inhibitory concentration of artesunate is observed when paracetamol is added to parasites in culture. We will investigate whether this effect is dependent on the infecting P. falciparum parasite strain
Paracetamol pharmacokinetics | 72 hours
  Pharmacokinetic modelling of oral paracetamol in severe and moderately severe malaria
Paracetamol pharmacodynamics | 72 hours
  Pharmacodynamics on variables including temperature and parasitemia.
Area under the plasma concentration versus time curve (AUC) | 72 hours
  for paracetamol
The maximum concentration (Cmax) | 72 hours
  for paracetamol

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Plewes, MD, Principal Investigator — University of Oxford
Locations (2):
- Bangladesh (2):
  - Chittagong Medical College Hospital, Chittagong
  - Ramu Upazilla Health Complex, Rāmu

REFERENCES:
- [Derived] Plewes K, Kingston HWF, Ghose A, Wattanakul T, Hassan MMU, Haider MS, Dutta PK, Islam MA, Alam S, Jahangir SM, Zahed ASM, Sattar MA, Chowdhury MAH, Herdman MT, Leopold SJ, Ishioka H, Piera KA, Charunwatthana P, Silamut K, Yeo TW, Lee SJ, Mukaka M, Maude RJ, Turner GDH, Faiz MA, Tarning J, Oates JA, Anstey NM, White NJ, Day NPJ, Hossain MA, Roberts Ii LJ, Dondorp AM. Acetaminophen as a Renoprotective Adjunctive Treatment in Patients With Severe and Moderately Severe Falciparum Malaria: A Randomized, Controlled, Open-Label Trial. Clin Infect Dis. 2018 Sep 14;67(7):991-999. doi: 10.1093/cid/ciy213. PMID 29538635